CLINICAL TRIAL: NCT03823157
Title: Tai Chi and eCB in Postmenopausal Women
Brief Title: Tai Chi and eCB in Women
Acronym: TC-eCB
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Tai Chi and eCB in women
Record Dates: First submitted 2019-01-28; First posted 2019-01-30 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Mind-body Exercise
MeSH Terms: interventions — Tai Ji

STUDY DESIGN:
Intervention Model Description: Tai Chi exercise
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tai Chi (Experimental): Tai Chi exercise
  Interventions: Behavioral: Tai Chi

INTERVENTIONS:
Behavioral: Tai Chi — mind-body exercise

SUMMARY:
The endocannabinoid system (ECS) is widely found in central and peripheral systems, and the immune system. Moderate-intensity aerobic exercise has shown to increase circulatory endocannabinoids. In this study, we will study Tai Chi, a mind-body moderate-intensity exercise, intervention for its effects on ECS in women. A pre-post design trial will be conducted on 18 qualified subjects. We will measure plasma eCB levels at baseline, before and after 4th session of Tai Chi. All data will be analyzed statistically at p<0.05.

DETAILED DESCRIPTION:
The endocannabinoid system (ECS) is widely found in central and peripheral systems, and the immune system. Emerging studies have shown endocannabinoid plays a role in appetite, pain sensation, control of chronic pain, macronutrient metabolism, mood/mood disorder, and regulation of immune cell functions. Moderate-intensity aerobic exercise has shown to increase circulatory endocannabinoids. Moderate-intensity exercise improves cognition, memory, and wellbeing in adults. Exercisers experience decreased tension, depression, and anger. Therefore, these findings in humans suggest a likely relationship for exercise effecting well-being via ECS. In this study, we will study Tai Chi, a mind-body moderate-intensity exercise, intervention for its effects on ECS in women. A pre-post design trial will be conducted on 15 qualified subjects. All subjects will be assigned to Tai Chi group for one week including 3 sessions, 60 minutes per session, on 3 non-consecutive days. We will measure plasma eCB levels at baseline, before and after 4th session of Tai Chi. All data will be analyzed statistically at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Postmenopausal women (menopause is defined as the absence of menstrual period for 12 months, not related to pregnancy/lactation, hormonal contraception). Age 40-70 years old with BMI between 25-35 kg/m2.
2. English literacy.

Exclusion Criteria:

1. prior experience with mind-body practice (e.g., TC, Qi Gong, yoga, meditation).
2. Severe medical limitations (i.e., dementia, symptomatic heart or vascular disease, or recent stroke) precluding full participation.
3. Medical/neurologic or other systemic diseases affecting the musculoskeletal systems (i.e. polio/Parkinson's/ multiple sclerosis, etc. in addition to cerebral vascular accident or stroke) and diabetes with peripheral neuropathy affecting their sensory/balance.
4. taking pain/anti-inflammatory and sleep medications within the 3 months before study starts.
5. taking hormone-replacement therapy within the 3 months before study starts.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 18 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
plasma eCB level | 1 week
  AEA and 2-AG

CONTACTS AND LOCATIONS:
Overall Officials: Chwan-li Shen, PhD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (1):
- Texas Tech University Health Sciences Center, Lubbock, Texas, United States